CLINICAL TRIAL: NCT00309439
Title: Studies of Serum PSA to Help Resolve the Current Implication of Alpha-linolenic Acid (ALA) and Prostate Cancer
Brief Title: ALA and Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: REB15636
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation; Diet Therapy; Prostate Cancer
MeSH Terms: conditions — Atrial Fibrillation; Prostatic Neoplasms

INTERVENTIONS:
Procedure: ALA-rich diet

SUMMARY:
The problem is the lack of data from randomized controlled trials to throw light on the ALA-prostate cancer issue. There is therefore a need to acquire evidence from a randomized controlled study to illustrate the effect of ALA on a surrogate marker for prostate cancer, namely prostate specific antigen (PSA). Demonstration that atrial fibrillation recurrence was reduced after cardioversion and that there was no adverse effect of 1 years of ALA feeding on PSA would go a considerable way to providing the required evidence that ALA in the human diet has no adverse effect on the prostate and so allow its use for cardiovascular risk reduction. hypothesis: The effect of ALA on PSA levels over time will be no different from the control, so providing supportive data for the view that ALA is not cancer promoting.

DETAILED DESCRIPTION:
In addition disturbing news on alpha-linolenic acid (ALA) has recently been reviewed by Brouwer and colleagues (J Nutr:2004). Their analyses suggests that ALA, as found in canola oil and other healthy foods, may cause prostate cancer even though there is good evidence that canola oil will prevent heart disease. This issue urgently needs further research.

In studies largely from the Harvard group, but suggested by additional studies from Uruguay and Spain, a link has been identified between ALA intake and prostate cancer. The Harvard studies are cohort studies where groups of approximately 40,000 doctors or health professionals have been followed up for periods of 10 years and the dietary intakes of ALA related to the subsequent development of aggressive prostate cancer. It must be stressed that these are not randomized crossover studies which are the currently accepted gold standard for evidence-based medicine and regulatory decision making. Nevertheless they raise concern over the health profile of a fatty acid with a growing reputation for cardiovascular disease prevention and a component of other healthy foods such as walnuts, flax, canola and soy.

The same Harvard group identified the deleterious effects on cardiovascular health of trans fatty acids in their cohort studies and this has resulted in a major effort to remove trans fatty acids from the food supply. On the other hand their identification of the benefits of vitamin E in their cohort studies has not been confirmed by subsequent randomized controlled trials. Although Dr Willett, the senior member of the Harvard group, has drawn surprisingly little attention to the negative findings with ALA, it remains a sticking point with regulators in the current debate over the inclusion and use of ALA in the food supply. This concern has been sufficient for the Natural Health Products Directorate of Health Canada to ask for a full proposal from us before we start studies on ALA in the prevention of atrial fibrillation due the apparently negative impact of ALA consumption on prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Blood samples available from Bordeaux

Exclusion Criteria:

* Blood samples not received from Bordeaux

Ages: 18 Years to 77 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, Principal Investigator — University of Toronto